CLINICAL TRIAL: NCT01691443
Title: Preliminary Study of the Substitution of Sensory Deficits of the Hand by a Medical Device Embedded : a Functional Assessment of Vibration Feedback on the Gripping Pressure in the Territory of the Median Nerve.
Brief Title: Functional Assessment of a Vibration Feedback on the Gripping Pressure in the Territory of the Median Nerve
Acronym: TEXIGLOVE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical problem with one of the medical device used for the study.
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Principal Investigator, AdministrateurCIC, principal investigator, University Hospital, Grenoble
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: DCIC 11 17; 2012-A00457-36 (Other: IDRCB)
Record Dates: First submitted 2012-07-12; First posted 2012-09-24 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Sensory Deficit

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Use of the glove (Experimental): The subject wear the glove for the time of the trial
  Interventions: Procedure: pressure sensor and wrist shaker, not marked CE, developped by Texisense

INTERVENTIONS:
Procedure: pressure sensor and wrist shaker, not marked CE, developped by Texisense

SUMMARY:
The objective of this study is to investigate the effect of vibration feedback on the gripping pressure in the territory of the median nerve.

ELIGIBILITY:
Inclusion Criteria:

* person between 18 and 45 years old
* affiliation to the french social security system or equivalent
* person signed a consent to participate
* for the patient group: person with post-traumatic sensory deficit in the territory of the right median nerve above the wrist (<S3 according Zachary modified Dellon).

Exclusion Criteria:

* person with a cognitive pathology incompatible with the use of the device, understanding and implementation of the protocol
* person with a concomitant nerve injury of any other nerve territory,
* person with pain or stiffness inconsistent with the achievement tests
* person with an allergy to any component of the device: polyamide, cotton, nickel, textile glue, rubber, plastic or latex,
* person with an infectious disease or dermatology of the right hand
* person deprived of freedom by judicial or administrative decision
* person hospitalized without their consent
* person under legal protection
* person hospitalized for psychiatric care
* pregnant and parturient women

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
intra-and inter-individual variance in pressure. | one year
  pressures are recorded during a test clamping with and without vibration feedback for the entire population

CONTACTS AND LOCATIONS:
Overall Officials: Denis Corcella, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Department of Plastic Surgery of the Hand and Burned - University Hospital Grenoble, Grenoble, France

REFERENCES:
- See also: Related Info — http://www.CIC-IT-grenoble.fr